CLINICAL TRIAL: NCT03885336
Title: Interpersonal Mechanisms of Smoking Relapse in Romantic Couples
Brief Title: Couples Dynamics and Smoking Cessation
Acronym: SCOR
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Matthew Kirkpatrick, Assistant Professor, University of Southern California
Other Study IDs: HS-16-00898
Record Dates: First submitted 2019-03-06; First posted 2019-03-21 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Smoking; Smoking Cessation; Cessation, Smoking; Smoking Behaviors; Smoking, Cigarette
MeSH Terms: conditions — Smoking; Smoking Cessation; Cigarette Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Both-Quit Group: Couples in which both individuals smoke and both individuals would like to quit smoking.
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — There are no interventions in this study. Participants are observed.

SUMMARY:
This study is about investigating smoking and attempts to quit smoking in couples. Participation will help determine better treatment efforts for couples who want to quit smoking. All study procedures will be conducted remotely, allowing couples to interact with study personnel through zoom.

ELIGIBILITY:
Inclusion Criteria:

* Couples must be in a relationship for more than 6 months with no plans to separate or move in the next 30 days.
* Participants must smoke at least 5 cigarettes per day for at least the past 2 years.

Exclusion Criteria:

* English non-fluency.
* Currently pregnant, nursing, or intend to become pregnant within the next 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants may live through the United States.
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2018-08-26 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Cigarette Craving | Throughout study completion, an average of 28 days
  This measure is obtained through the completion of the Brief Questionnaire of Smoking Urges.
Confidence in Quit Attempt | Throughout study completion, an average of 28 days
  This measure is obtained through the completion of the Abstinence Self-Efficacy Questionnaire.
Mood | Throughout study completion, an average of 28 days
  This measure is obtained through the completion of the Profile of Mood States Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kirkpatrick, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No